CLINICAL TRIAL: NCT02266667
Title: Evaluation of the Efficiency of Nemost Growing Spine Device Associated With Physiotherapy in the Surgical Treatment of Progressive Scoliosis of the Child
Brief Title: Surgical Treatment of Progressive Scoliosis With "NEMOST" Growing Rod
Acronym: NEMOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Company EUROS (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P140301
Record Dates: First submitted 2014-07-25; First posted 2014-10-17 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Progressive Scoliosis
Keywords: NEMOT device; pediatrics; surgery; progressive scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive scoliosis (Experimental): Children with progressive scoliosis
  Interventions: Device: 1 NEMOST rod :unilateral vertebral-pelvic implantation
- Neuromuscular scoliosis (Experimental): Children with neuromuscular scoliosis
  Interventions: Device: 2 NEMOST rods : bilateral vertebral-pelvic implantation

INTERVENTIONS:
Device: 2 NEMOST rods : bilateral vertebral-pelvic implantation — Implantation of two NEMOST rods (bilateral vertebral-pelvic implantation)
  Arms: Neuromuscular scoliosis
Device: 1 NEMOST rod :unilateral vertebral-pelvic implantation — Implantation of one NEMOST rod (unilateral vertebral-pelvic implantation)
  Arms: Progressive scoliosis

SUMMARY:
The purpose of this study is to evaluate the performance of the device "NEMOST" on maintaining of the correction of the scoliosis with growth preservation and avoiding iterative surgeries.

Objective of this study is to evaluate the performance of the growing device "NEMOST" associated to physiotherapy at 12 months postoperatively in patients treated for progressive scoliosis and to evaluate its safety.

DETAILED DESCRIPTION:
A number of scoliosis in the child remain progressive despite conservative treatment well conducted. Nowadays the most used treatment is early surgical treatment by the spinal instrumentation without graft called "growing rods". The use of growing rods in patients with progressive scoliosis requires several repeated surgeries (every 6 to 12 months) in order to follow the growth of children. These repeated surgeries lead to a significant increased risk of complications, that's why many teams around the world have been seeking solutions which allow to obtain a rod expansion without repeated surgery.

The purpose of our study is the evaluation of the use of medical device that will perform the correction of scoliosis and, at the same time, preserve the growth of the child's spine. In addition, the purpose of clinical investigation is to test the theory that distraction effort may be exercised without surgery thanks to traction manoeuvres and physiotherapy. This could allow to obtain in patients with progressive scoliosis, correction of spinal deformity while avoiding many repeated surgeries. Our reference device is growing rod "NEMOST". When implanted, NEMOST rod is immediately turned on, for correcting and maintaining the correction of spinal deformity. After implantation, depending on development in Cobb angle, one or more elongations can be made by sliding the notched portion of the rod in its tunnel by a distraction effort (traction equipments and physiotherapy).

Therefore, the growth device NEMOST will allow to continue, on request, the correction of spinal deformity by performing a distraction by external manoeuvres on the notched part without the need for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 5 to 15 years old
* Patient with neuromuscular scoliosis or progressive scoliosis resistant to conservative treatment
* Patient with an indication of first-line surgery without graft
* Patient with low skeletal maturity (Risser test = 0 and triradiate growth cartilages still open)
* Signing of the consent by the holder (s) of parental authority and the investigator
* Affiliated patient to a health service or entitled patient

Exclusion Criteria:

* Patient with a history of spinal surgery
* Patient weighing more than 30 kg and with progressive scoliosis other than neuromuscular
* Patient with contra-indication to Nemost device, that is to say:

  * Inflammation or acute Infection, local or systemic,
  * Allergy or intolerance titanium or polyetheretherketone,
  * Pathology or poor bone quality might compromise the attachment of the device,
  * Nonreducible Scoliosis,
  * Skin Substance insufficient to cover the wound,
  * Pathological Obesity,
  * Fracture and / or spinal tumor,
  * Patient whose behavior presents a risk of failure for the device.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
No surgical reoperation | 12 months
  The lack of indication of surgical reoperations means that the correction of scoliosis is satisfactory and the growth had been maintained
No worsening of Cobb angle by more than 15 degrees since the initial correction | 12 months
  A worsening of the Cobb angle by more than 15 ° since the initial correction is considered an indication of reoperation

SECONDARY OUTCOMES:
Cobb angle | 3 months
  Radiographic measure : less than 15 degrees since the initial correction
Cobb angle | 6 months
  Radiographic measure : less than 15 degrees since the initial correction
Cobb angle (degree) | 18 months
  Radiographic measure : less than 15 degrees since the initial correction
reserve rod (mm) | 3 months
  This amount reflects the actual elongation of the device
reserve rod (mm) | 6 months
  This amount reflects the actual elongation of the device
reserve rod (mm) | 12 months
  This amount reflects the actual elongation of the device
reserve rod (mm) | 18 months
  This amount reflects the actual elongation of the device
T1-T12 segment and T1-S1 segment | 3 months
  which reflect the real growth of the spine
T1-T12 segment and T1-S1 segment | 6 months
  which reflect the real growth of the spine
T1-T12 segment and T1-S1 segment | 12 months
  which reflect the real growth of the spine
T1-T12 segment and T1-S1 segment | 18 months
  which reflect the real growth of the spine
respiratory function | 6 months
  Translated chest and lung growth, as well as the actual improvement of respiratory function
respiratory function | 12 months
  Translated chest and lung growth, as well as the actual improvement of respiratory function
respiratory function | 18 months
  Translated chest and lung growth, as well as the actual improvement of respiratory function
Pelvic obliquity (mm) | 3 months
  translated improving the overall balance of the trunk of the patient for the group of children with neuromuscular scoliosis
Pelvic obliquity (mm) | 6 months
  translated improving the overall balance of the trunk of the patient for the group of children with neuromuscular scoliosis
Pelvic obliquity (mm) | 12 months
  translated improving the overall balance of the trunk of the patient for the group of children with neuromuscular scoliosis
Pelvic obliquity (mm) | 18 months
  translated improving the overall balance of the trunk of the patient for the group of children with neuromuscular scoliosis
Safety of NEMOST | 3 months
  Nature-incidence and severity of complications due to NEMOST : infections, elongation failure, problems with healing after surgery, neurological deficit) Nature and incidence of any medical and surgical intervention in relation to device NEMOST
Safety of NEMOST | 6 months
  Nature-incidence and severity of complications due to NEMOST : infections, elongation failure, problems with healing after surgery, neurological deficit) Nature and incidence of any medical and surgical intervention in relation to device NEMOST
Safety of NEMOST | 12 months
  Nature-incidence and severity of complications due to NEMOST : infections, elongation failure, problems with healing after surgery, neurological deficit) Nature and incidence of any medical and surgical intervention in relation to device NEMOST
Safety of NEMOST | 18 months
  Nature-incidence and severity of complications due to NEMOST : infections, elongation failure, problems with healing after surgery, neurological deficit) Nature and incidence of any medical and surgical intervention in relation to device NEMOST
Weight (kg) | Every month for 18 months
  Reflecting the improvement in the general and trophic status of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Nejib KHOURI, MD, PhD, Study Director — Hospital Necker Enfants Malades
Locations (1):
- Hospital Necker Enfants Malades, Paris, France

REFERENCES:
- [Background] Miladi L, Khouri N, Pradon J, Elie C, Treluyer JM. One-way self-expanding rod for early-onset scoliosis: early results of a clinical trial of 20 patients. Eur Spine J. 2021 Mar;30(3):749-758. doi: 10.1007/s00586-021-06732-4. Epub 2021 Jan 24. PMID 33486593